CLINICAL TRIAL: NCT07385638
Title: Phase 2, Open-label Evaluation of Olorofim in Early Coccidioidal Meningitis
Brief Title: Olorofim in Early Coccidioidal Meningitis
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fariba Donovan (Other)
Collaborators: F2G Biotech GmbH (Industry)
Responsible Party: Sponsor-Investigator, Fariba Donovan, MD, PhD, University of Arizona
Organization: University of Arizona (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Study 00006853
Record Dates: First submitted 2026-01-23; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Coccidioidal Meningitis
Keywords: coccidioidomycosis
MeSH Terms: conditions — Coccidioidal Meningitis; Coccidioidomycosis | interventions — olorofim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- olorofim (Experimental): Participants will receive treatment with olorofim
  Interventions: Drug: olorofim

INTERVENTIONS:
Drug: olorofim — Single group study - all participants will receive olorofim treatment

SUMMARY:
This research study is being conducted to learn more about the use of olorofim in Coccidioidal (Cocci) meningitis, a rare but serious fungal infection that affects the brain and spinal cord. The study is exploratory, meaning that early information is being gathered to better understand the effectiveness of olorofim in coccidioidal meningitis in its early stages. The study plans to enroll approximately 10 to 12 participants who have been recently diagnosed-within the last 4 to 8 weeks-and who do not have a ventriculoperitoneal (VP) shunt, a medical device sometimes used to relieve pressure in the brain. Participants will be followed for approximately 6 months, during which health information will be collected to evaluate disease progression and response to treatment. Participants may have the opportunity to enroll in the olorofim Managed Access Program to continue treatment after completion of the study period.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients aged ≥ 18 years and weighing ≥ 40 kg, able to understand and consent in English, who have been fully informed and:

   a) who have given voluntary written informed consent, or whose legally authorized representative(s) has been fully informed and has given voluntary written informed consent if applicable, and in compliance with local regulations OR
2. b) who have given oral informed consent witnessed in writing by an independent person and in compliance with local regulations for patients who are unable to write and/or read but who fully understand the oral information given by the Investigator (or nominated representative).
3. Ongoing coccidioidomycotic meningitis diagnosed within 8 weeks prior to enrolment.
4. Ongoing symptoms due to coccidioidomycosis are such that the risk-benefit of treatment with an investigational agent with a hepatic signal requiring careful monitoring is judged favorable based on meeting criteria
5. Female patients must be non-lactating and at no risk of pregnancy for one of the following reasons:

   * Postmenopausal for at least 1 year;
   * Post-hysterectomy and/or post-bilateral oophorectomy;
   * Of childbearing potential, with a negative urine or serum human chorionic gonadotropin pregnancy test at the screening visit and must be using one of listed below highly effective method of birth control throughout the course of the study period and up to and including 30 days after stopping study drug

     * Established use of oral, injected, transdermal, intravaginal, or implanted hormonal methods of contraception associated with inhibition of ovulation
     * Placement of an intrauterine device or intrauterine hormone-releasing system
     * Male sterilization
     * Bilateral tubal occlusion
     * Sexual abstinence (reliable sexual abstinence is acceptable but periodic abstinence [e.g., calendar, ovulation, symptom-thermal, or post-ovulation methods] and withdrawal are not acceptable).
6. Male patients with female partners of childbearing potential must either totally abstain from sexual intercourse or use a highly effective means of contraception throughout study participation and agree to continue its use for 30 days after stopping study drug and may not donate semen during this time.

Exclusion Criteria:

1. Patients who are unconscious.
2. Patients who are pregnant or breastfeeding.
3. Known history of allergy, hypersensitivity, or any serious reaction to any component of the olorofim.
4. Patients with or planned placement of indwelling CNS hardware (e.g. reservoirs, shunts, ventriculostomies, or external drainage tubes).
5. Patients with a second fungal infection requiring systemic antifungal treatment or prophylaxis, other than Pneumocystis jirovecii infections and cutaneous fungal infections treated topically.
6. Patients with microbiological findings (e.g., bacteriological, virological) or other potential conditions that are temporally related and suggest a different than study indication etiology.
7. HIV infection but not currently receiving antiretroviral therapy. In cases where HIV infection is first diagnosed at the same time as the invasive fungal infection, if antiretroviral therapy is commenced at the time of enrollment, then such patients are eligible for enrolment
8. Any known or suspected medical condition or social circumstance of the patient that may jeopardize adherence to the protocol requirements or impede the accurate measurement of efficacy.
9. Patients with a concomitant medical condition that, in the opinion of the Investigator, may be an unacceptable additional risk to the patient should he/she participate in the study.
10. Patients who have received prior treatment with olorofim/F901318.
11. Treatment with any investigational drug within the 30 days prior to the first administration of study drug except for unblinded protocols (eg, open-label oncological regimen variations or biologic studies). Prior to enrolling patients who are on other open-label studies, it is the site's responsibility to ensure that the study criteria for that study allow for enrollment into this study.
12. Patients receiving treatment limited to supportive care due to predicted short survival time.
13. Patients with a baseline prolongation of QT using Fridericia's Correction Formula (QTcF) ≥ 500 msec, or at high risk for QT/QTc prolongation, eg,

    1. A family history of long QT syndrome
    2. Other known pro-arrhythmic conditions
    3. Risk factors for Torsade de Pointes (e.g., uncompensated heart failure, abnormal plasma potassium or magnesium levels that cannot be corrected, an unstable cardiac condition during the last 30 days).
14. Evidence of hepatic dysfunction with any of the following abnormal laboratory parameters at screening:

    1. Total bilirubin ≥ 2 × upper limit of the normal range (ULN), OR
    2. Alanine transaminase (ALT) or aspartate transaminase (AST) ≥ 3 × ULN, OR
    3. Patients with known cirrhosis or chronic hepatic failure (regardless of ALT/AST/total bilirubin).

    Liver transplant recipients may be enrolled if their laboratory parameters do not meet the laboratory exclusions given above.
15. Prohibited concomitant medications. Concomitant administration of inhibitors of human dihydro-orotate dehydrogenase (DHODH), teriflunomide, leflunomide, and systemic use of cannabis/cannabinoid preparations, including tetrahydrocannabinol (THC) and cannabidiol (CBD) are prohibited. There are currently no other absolutely prohibited concomitant medications for olorofim but there are medications with potentially significant drug-drug interactions (DDIs) with olorofim or SOC and the management of potential interactions should be considered before study enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2026-03-15 (Estimated); Primary Completion 2027-03-15 (Estimated); Study Completion 2027-06-15 (Estimated)

PRIMARY OUTCOMES:
Safety: Number of participants with ≥1 treatment-emergent adverse event | First dose through end of treatment and 4-week follow-up
  Counts and proportions of participants experiencing at least one adverse event after initiation of olorofim, regardless of causality. Adverse events will be coded and graded according to CTCAE v5.0.

SECONDARY OUTCOMES:
Efficacy: Investigator-assessed clinical response over 24 weeks | Baseline through Week 24 (End of Treatment)
  Proportion of participants with improvement or resolution of coccidioidal meningitis-related clinical signs and symptoms compared with baseline, as assessed by the investigator at protocol-specified visits.
Efficacy: Change from baseline in Coccidioides serum complement fixation titers | Baseline through Week 24
  Change in serum complement fixation titers from baseline, measured at scheduled study visits, as an indicator of mycological and disease response.
Efficacy: Radiological response assessed by imaging | Baseline through Week 24
  Proportion of participants with stable or improved radiological findings related to coccidioidal meningitis on clinically indicated imaging studies compared with baseline.
Efficacy: Investigator-assessed overall treatment response | Baseline through Week 24
  Proportion of participants with overall response based on integration of clinical status, radiological findings (if available), and mycological/serologic data, as assessed by the investigator using protocol-defined criteria.
Efficacy: All-cause mortality | Baseline through Week 24 and 4-week follow-up
  Proportion of participants who die from any cause during treatment or follow-up.
Patient-reported Outcome: Change from baseline in Modified Zubrod Performance Score | Baseline through Week 24
  Change from baseline in MZ-PS, a measure of functional performance status.
Patient-reported Outcome: Change from baseline in Valley Fever Patient-Reported Outcomes (VF-PRO) score | Baseline through Week 24
  Change from baseline in VF-PRO questionnaire scores assessing symptom burden and quality of life related to coccidioidomycosis.
Patient-reported Outcome: Change from baseline in Clinical Global Impression-Severity (CGI-S) and Patient Global Impression-Severity (PGI-S) | Baseline through Week 24
  Change from baseline in investigator-rated (CGI-S) and patient-reported (PGI-S) disease severity scores. (separate scales but reported similarly)
ECG Sub-Study: Change from baseline in QTcF interval | Day 10-21 (single study day)
  Change in QT interval corrected using Fridericia's formula (QTcF), measured using continuous Holter ECG monitoring and time-matched with plasma olorofim concentrations in a subset of participants.

CONTACTS AND LOCATIONS:
Overall Officials: Fariba Donovan, MD, PhD, Principal Investigator — University of Arizona
Locations (1):
- Banner University Medical Center, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD), including the analyzable dataset and associated metadata, will be shared with the study collaborator, F2G Ltd., for purposes of regulatory support, safety evaluation, and further analysis related to olorofim. Data shared will not include direct identifiers and will be coded prior to transfer.
Supporting Information: CSR
Access Criteria: Access to the de-identified IPD will be limited to F2G Ltd. and authorized third-party vendors acting on behalf of the collaborator, under data use agreements that specify permitted uses and prohibit re-identification. Data will not be made publicly available. Study results may be disseminated through scientific publications and presentations.